CLINICAL TRIAL: NCT02693210
Title: A Randomised, Double Dummy Controlled, Parallel Group Study of the Efficacy and Safety of MabThera (Rituximab) Alone or in Combination With Either Cyclophosphamide or Methotrexate, in Patients With Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Mabthera Alone and in Combination With Either Cyclophosphamide or Methotrexate in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA16291
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cyclophosphamide; Methotrexate; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group A: Methotrexate (Active Comparator): Participants will receive methotrexate at dosage >=10 milligrams per week (mg/week) orally as determined by the investigator. They also receive placebo infusion on days 1 and 15 in place of rituximab and on Days 3 and 17 in place of cyclophosphamide.
  Interventions: Drug: Methotrexate; Other: Placebo Cyclophosphamide; Other: Placebo Rituximab
- Group B: Rituximab Monotherapy (Experimental): Participants will receive 1 g intravenous infusions of rituximab on Days 1 and 15. They also receive Weekly placebo orally instead of methotrexate and placebo infusion in place of cyclophosphamide on Days 3 and 17.
  Interventions: Other: Placebo Cyclophosphamide; Other: Placebo Methotrexate; Drug: Rituximab
- Group C: Rituximab and Cyclophosphamide (Experimental): Participants will receive 1g IV infusion of rituximab on Days 1 and 15 and 750 mg infusion of Cyclophosphamide on Days 3 and 17. They also receive weekly oral placebo in place of methotrexate.
  Interventions: Drug: Cyclophosphamide; Other: Placebo Methotrexate; Drug: Rituximab
- Group D: Methotrexate and Rituximab (Experimental): Participants will receive >=10 mg/week methotrexate orally along with 2 times 1 gram (g) rituximab IV infusions on Days 1 and 15. Participants will also receive placebo infusions on Days 3 and 17 in place of cyclophosphamide.
  Interventions: Drug: Methotrexate; Other: Placebo Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Participants will receive 750 mg infusions of cyclophosphamide on Days 3 and 17
  Arms: Group C: Rituximab and Cyclophosphamide
Drug: Methotrexate — Participants will receive >= 10 mg/week methotrexate orally up to 24 weeks
  Arms: Group A: Methotrexate; Group D: Methotrexate and Rituximab
Other: Placebo Cyclophosphamide — Participants will receive placebo in place of cyclophosphamide on Days 3 and 17
  Arms: Group A: Methotrexate; Group B: Rituximab Monotherapy; Group D: Methotrexate and Rituximab
Other: Placebo Methotrexate — Participants will receive weekly oral placebo in place of Methotrexate
  Arms: Group B: Rituximab Monotherapy; Group C: Rituximab and Cyclophosphamide
Other: Placebo Rituximab — Participants will receive placebo in place of rituximab on days 1 and 15
  Arms: Group A: Methotrexate
Drug: Rituximab — Participants will receive 1g infusions of rituximab on Days 1 and 15
  Arms: Group B: Rituximab Monotherapy; Group C: Rituximab and Cyclophosphamide; Group D: Methotrexate and Rituximab

SUMMARY:
WA16291 is a Phase IIa "proof-of-concept" study. The primary objective of this study is to determine the safety and efficacy of rituximab (a B cell depleting chimeric monoclonal antibody) used either as monotherapy or in combination with methotrexate or cyclophosphamide in participants with rheumatoid arthritis who have failed prior Disease Modifying Anti-Rheumatic Drug (DMARD) therapy and currently have an inadequate clinical response to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe rheumatoid arthritis (RA) who have previously failed 1-5 DMARDS who currently have partial clinical response to treatment with methotrexate
* Using methotrexate as a single DMARD for at least 16 weeks, of which the last 4 weeks prior to baseline on a stable oral dose greater than or equal to (>=) 10 milligrams per week (mg/week)
* >=21 years of age
* Swollen Joint Count (SJC) and Tender Joint Count (TJC) >= 8 (out of 66 and 68 joints respectively)
* At least 2 of the following parameters at Baseline: C- Reactive Protein >= 15 mg/dL; Erythrocyte Sedimentation Rate >= 30 millimeters per hour (mm/hr); Morning stiffness >45 minutes
* Rheumatoid factor titer >=20 International units per milliliter (IU/mL)
* Corticosteroid (less than or equal to [=<] 12.5 milligrams per deciliter [mg/d] prednisone or equivalent) or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) are permitted if stable for at least 4 weeks prior to baseline

Exclusion Criteria:

* American Rheumatism Association (ARA) Class IV RA disease
* Concurrent treatment with any DMARD (apart from randomized treatment) or anti-TNF-alpha therapy
* Active infection or history of recurrent significant infection
* Prior history of cancer including solid tumors and hematologic malignancies (except basal carcinoma of the skin that have been excised and cured)
* Evidence of serious uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders
* Bone/joint surgery within 6 weeks prior to screening
* Rheumatic Autoimmune disease other than RA
* Active rheumatoid vasculitis
* Prior history of gout
* Chronic fatigue syndrome

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2001-02; Primary Completion 2002-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving American College of Rheumatology (ACR) 50 response at Week 24 | Week 24

SECONDARY OUTCOMES:
Percentage of participants achieving ACR 20 and ACR 70 responses at Week 24 | Week 24
Area Under the Curve (AUC) of American College of Rheumatology Response (ACRn) | Baseline up to Week 24
AUC of the mean Disease Activity Scores (DAS) | Baseline up to Week 24
Change from Baseline in the Swollen Joint Count | Baseline, Weeks 12, 16, 20 and 24
Change from Baseline in the Tender Joint Count | Baseline, Weeks 12, 16, 20 and 24
Change from Baseline in participant's global assessment of disease activity using a Visual Analog Scale (VAS) | Baseline, Weeks 8, 12, 16, 20 and 24
Change from Baseline in physician's global assessment of disease activity using VAS | Baseline, Weeks 8, 12, 16, 20 and 24
Change from Baseline in the Health Assessment Questionnaire - Disease Index (HAQ-DI) scores | Baseline, Weeks 12, 16, 20 and 24
Change from Baseline in participant's pain measured by VAS | Baseline, Weeks 12, 16, 20 and 24
Change from Baseline in C-Reactive Protein (CRP) Levels | Baseline, Weeks 12, 16, 20 and 24
Change from Baseline in Erythrocyte Sedimentation Rate (ESR) | Baseline, Weeks 12, 16, 20 and 24
Mean change in Rheumatoid factor levels at 24 weeks | Baseline and Week 24
Percentage of participants who withdrew due to insufficient therapeutic response | Up to 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hofffmann-La Roche
Locations (31):
- Australia (3):
  - Darlinghurst
  - Kogarah
  - Woodville
- Belgium (3):
  - Diepenbeek
  - Ghent
  - Liège
- Canada (3):
  - Winnipeg, Manitoba
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- Germany (3):
  - Leipzig
  - Ratingen
  - Wiesbaden
- Haifa, Israel
- Italy (4):
  - Brescia
  - Genova
  - Modena
  - Siena
- Leiden, Netherlands
- Poland (4):
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Spain (4):
  - Guadalajara
  - Madrid
  - San Cristóbal de La Laguna
  - Seville
- United Kingdom (4):
  - Cannock
  - Leeds
  - London
  - Stoke-on-Trent